CLINICAL TRIAL: NCT05460845
Title: Low-Carbohydrate Diet to Reduce Pain and Increase Quality of Life in Amputees
Brief Title: The Pain in Amputees Reduced by Administration of Diet Examination
Acronym: PARADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Robert Sorge, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300008971
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Amputation; Phantom Limb Pain; Residual Limb Pain
MeSH Terms: conditions — Phantom Limb | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase 2 Intervention (Experimental): Low-Carbohydrate Diet
  Interventions: Behavioral: Low-Carbohydrate Diet

INTERVENTIONS:
Behavioral: Low-Carbohydrate Diet — Using a meal delivery service and a list of prepared meals and recipes, foods/meals will be delivered to participants weekly to maintain daily net carbohydrate intake to less than 40 grams.
  Other Names: LCD

SUMMARY:
Phantom limb pain (PLP) is defined as pain or discomfort in a missing limb following amputation, whereas residual limb pain (RLP) is often experienced as pain at the site of amputation. Unfortunately, PLP can affect as many as 80% of upper- or lower-extremity amputees, with 40-60% also experiencing RLP. There are many theories regarding the mechanisms underlying these types of pain, but effective treatments remain elusive .Amputation of a limb is often accompanied by a traumatic event that can be emotionally devastating. Consequently, studies have reported high levels of depression in this population, up to 80%. Other studies have reported elevated levels of depression (70%), suicidality (30%) and posttraumatic stress disorder (PTSD, 20%) with PTSD being highly correlated with PLP. Thus, it is critical that effective treatments be employed that address, not only the chronic pain, but the comorbid conditions as well.

Diet interventions have been utilized as a non-pharmacological method to reduce pain and/or inflammation. We have shown that a low-carbohydrate diet (LCD) reduced pain independent of weight loss. Importantly, we observed a reduction in depressive symptomology and improved quality of life (QOL) following the LCD. Thus, it is reasonable to expect that the LCD may have beneficial effects of pain experience and also on measures of QOL.

Phase 1: To characterize the dietary habits, pain severity and psychological well-being of the local amputee population.

Hypotheses: We expect that the local population will show high prevalence of phantom limb pain (PLP) and/or residual limb pain (RLP). Self-report of depressive symptomology, poor-quality diet, will coincide with low QOL reports.

Phase 2: To assess the feasibility and efficacy of a low-carbohydrate diet (LCD) to reduce pain and increase QOL in amputees.

Hypotheses: All participants will complete the 6-week LCD. Compared to baseline, a 6-week LCD will reduce self-reports of pain and depressive symptoms. Overall QOL will improve over 6 weeks with concomitant improved mood and sleep.

DETAILED DESCRIPTION:
Phase 1: Baseline Demographics

Participants: We expect to recruit 40 participants (male or female, aged 18-65 years) for Phase 1. Inclusion criteria will be: PLP/RLP for at least 6 months (>4/10 on visual analogue scale), amputation at least 6 months prior. Exclusion criteria will include: inability to read/understand English, current infection at amputation site. We will collect clinical data related to amputation (cause, date, affected limb, level) and sociodemographic information (sex, gender, race, income, education, employment status etc.), in addition to a 24-hour diet recall to assess regular diet habits. Furthermore, we will collect the following:

Pain-Related Questionnaires: Chronic PLP/RLP will be assessed using the Brief Pain Inventory (BPI), Neuropathic Pain Questionnaire (NPQ), and the McGill Pain Questionnaire - Short Form (MPQ-SF). The BPI is used to assess the severity of pain and the degree to which that pain interferes with daily activities. This inventory also allows for reports on medications used to treat pain. The NPQ is specific to the type of pain commonly experienced in PLP/RLP, consisting of sensory, affective and sensitivity measures. The MPQ-SF is a standard metric whereby patients can select descriptors to categorize their pain experience more fully across sensory, affective, and evaluative dimensions.

QOL-Related Questionnaires: The Short-Form 36 (SF-36) measures general health status and quality of life across eight domains that are relevant to assessment of a diet intervention. Depression and mood will be assessed using the Center for Epidemiological Studies - Depression (CES-D) scale. The CES-D assesses depression as well as sleep, appetite and loneliness and can be used to identify those at risk for clinical depression (score >16). Higher scores indicate more depressive symptoms. We will utilize the Pittsburgh Sleep Quality Index (PSQI) to assess self-reported sleep. We believe that the LCD will increase restful sleep. The Nottingham Extended Activities of Daily Living Scale (NEADL) assesses regular household and leisure activities and has been used to measure QOL in amputees.

Psychological Questionnaires: The Acceptance and Action Questionnaire (AAQ) will be used to assess psychological flexibility. The Cognitive Flexibility Scale (CFS) will assess cognitive flexibility through ratings of agreement with 12 statements. The Multidimensional Psychological Flexibility Inventory (MPFI) will assess multiple domains of cognitive flexibility. The Pain Resilience Scale (PRS) will be used as a specific means to investigate resilience (behavioral perseverance and cognitive positivity) for those with chronic pain.

Phase 2: Diet Intervention

Participants: Following the collection of baseline demographic information at the Spain Amputee Clinic, we will recruit 10 individuals (male or female, aged 18-65 years) for our diet intervention phase. Inclusion criteria will be: PLP/RLP for at least 6 months (>4/10 on visual analogue scale), amputation at least 6 months prior. Exclusion criteria will include: inability to read/understand English, current infection at amputation site, unmedicated diabetes, unwillingness to follow prescribed diet, recent weight change (>4 kg in past month), currently on a diet, history of eating disorders or other psychiatric disorders requiring hospitalization within the past 6 months, digestive diseases, difficulty chewing or swallowing, reliance on others for meal preparation, cardiovascular or pulmonary disease, daily opioid pain medications, use of medications known to alter metabolism or digestion (e.g., proton-pump inhibitors), use of anti-hypertensive medications that affect glucose tolerance, participation in extreme exercise.

Diet Intervention: The LCD is designed to reduce daily intake of carbohydrates. Participants are directed to reduce their total (not net) carbohydrate intake to ≤ 40 g/day. Meals will be offered such that no combination of chosen meals will exceed our limit. Fats will not be restricted, nor will protein (meats, eggs). However, the provision of meals by our study personnel will allow us to cap the total proteins and fats, reducing this source of variability. Fruits will be restricted and vegetables permitted in limited quantities (2 cups/day of leafy greens, 1 cup/day non-starchy vegetables, etc.). Participants will be instructed as to the types and quantities of beverages that are permitted to accompany the LCD. Artificial carbohydrate-free sweeteners (stevia or sucralose) will be permitted, but powdered sweeteners (aspartame, saccharin, stevia, sucralose) can only be used in limited quantities as they contain maltodextrin (1 g of rapidly digesting carbohydrate). It is worth noting that our LCD is not directed at weight loss, but that we expect that some weight loss will occur.

Food Provision: Adherence to a LCD is associated with increased quality of life and decreased pain and disability. However, for a number of participants, diet prescriptions of any type are dramatic lifestyle changes that require oversight to maintain adherence. To overcome the difficulties in maintaining the assigned diets, food will be provided weekly using the Shipt service and local grocery stores. Participants will be given a list of available meals and will choose one week of meals (breakfast, lunch, dinner, snacks) in consultation with study personnel to increase adherence and contact time. This service will provide for greater control over the foods being consumed by the diet groups, though checklists will be required to document adherence and extra foods/beverages aside from the foods provided. Participants with persistent poor adherence will be counseled by study personnel and may be removed from the study.

Diet-Related Questionnaires: The short form of the Household Food Security Scale (HFSS-SF) will be used to assess food security. At baseline and every 3 weeks, participants will complete the modified Trait and State Food-Cravings Questionnaire, which is designed to assess hunger, cravings, and other measures associated with perception of ability to refrain from eating. At the end of Phase 2, participants will complete a modified version of the Treatment Satisfaction Questionnaire for Medication (TSQM) to assess attitudes and satisfaction regarding the dietary prescriptions provided and changes in overall health achieved.

Anthropometric Measures: Weight will be measured at every visit. The same calibrated scale will be used for all measurements. Height, waist circumference, heart rate and blood pressure will also be measured.

Statistical Analysis: Data collected in Phase 1 will be used to characterize levels of pain and other psychosocial outcome variables within this participant population. Descriptive statistics will be used to express these data. In Phase 2, feasibility will be determined by adherence and retention in the study. Preliminary efficacy will be detected by comparison of various outcome measures across time (baseline, weeks 3 and 6), using repeated measures analysis of variance. Consequently, we will have 80% power to detect an effect size of 0.44 with our alpha set to 0.05 for single measures outlined above (i.e., SF-36 scores, BPI scores, etc.). Due to the relatively small sample size and the nature of the pilot, we will not adjust for multiple comparisons.

Clinically-Meaningful Differences: Group mean differences are not always reflective of clinically-meaningful differences at the individual level. Therefore, an analysis will be carried out using published clinically-meaningful differences in baseline pain intensity score. Briefly, a reduction of ≥1.7 on an 11-point rating scale) is considered clinically-meaningful. In our feasibility trial, we saw that the LCD was more effective in improving pain, according to the criteria described above.

ELIGIBILITY:
Phase 1 Inclusion Criteria:

* Amputation at least 6 months prior

Phase 1 Exclusion Criteria:

* Inability to read/understand English
* Active infection at amputation site

Phase 2 Inclusion Criteria:

* PLP/RLP for at least 6 months (>4/10 on visual analogue scale)
* Amputation at least 6 months prior

Phase 2 Exclusion Criteria:

* Inability to read/understand English
* Current infection at amputation site
* Unmedicated diabetes
* Unwillingness to follow prescribed diet
* Recent weight change (>4 kg in past month)
* Currently on a prescribed diet or consuming less than 100 g of daily carbohydrates
* History of eating disorders or other psychiatric disorders requiring hospitalization within the past 6 months
* Digestive diseases
* Difficulty chewing or swallowing
* Reliance on others for meal preparation
* Uncontrolled cardiovascular or pulmonary disease
* Daily opioid pain medications
* Use of medications known to alter metabolism or digestion (e.g., proton-pump inhibitors)
* Use of anti-hypertensive medications that affect glucose tolerance
* Participation in extreme exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
BPI Pain Severity Change | Baseline (week 0), immediately after the intervention (week 6)
  BPI pain severity is an average score out of 10.
BPI Pain Interference Change | Baseline (week 0), immediately after the intervention (week 6)
  BPI pain interference is an average score from 9 items out of 10.
SF-36 overall score change | Baseline (week 0), immediately after the intervention (week 6)
  The Short Form 36 (SF-36) quality of life score is a 0-150 score with higher scores reflecting poorer quality of life. Scores in each of the 7 sections (general health, limitations, physical health, emotional health, social activities, pain and energy) are summed to provide an overall quality of life score. Change scores will be calculated.

SECONDARY OUTCOMES:
NPQ score change | Baseline (week 0), immediately after the intervention (week 6)
  The NPQ is specific to the type of pain commonly experienced in PLP/RLP, consisting of sensory, affective and sensitivity measures.
CES-D score change | Baseline (week 0), immediately after the intervention (week 6)
  The CES-D assesses depression as well as sleep, appetite and loneliness and can be used to identify those at risk for clinical depression (score >16). Higher scores indicate more depressive symptoms.
PSQI change score | Baseline (week 0), immediately after the intervention (week 6)
  The PSQI assesses sleep quality through self-report.
NEADL change score | Baseline (week 0), immediately after the intervention (week 6)
  The NEADL assesses regular household and leisure activities and has been used to measure QOL in amputees.
PROMIS-57 domain change | Baseline (week 0), immediately after the intervention (week 6)
  The PROMIS-57 will be used to assess many domains of QOL in Phase 1 and 2. For each domain, the raw scores will summated and adjusted using the T-score tables to provide standardized sores. These scores will be compared across time (Phase 2 only).
AAQ change score | Baseline (week 0), immediately after the intervention (week 6)
  The Acceptance and Action Questionnaire will be used to assess psychological flexibility in Phase 2. Scores will be summated and an average score calculated.
CFS score change | Baseline (week 0), immediately after the intervention (week 6)
  The Cognitive Flexibility Scale is a 12-item scale using a Likert model to identify the degree of agreement with 12 statements. Responses are summated.
MPFI score change | Baseline (week 0), immediately after the intervention (week 6)
  The Multidimensional Psychological Flexibility Inventory is another means to assess flexibility in thinking across 60 items and 6 dimensions of psychological flexibility. Responses are assigned values and each domain subscale is summated.
PRS total and subscale score change | Baseline (week 0), immediately after the intervention (week 6)
  The Pain Resilience Scale is a 14-item scale that assesses resilience in the presence of stressful or painful conditions and includes two subscales (behavioral perseverance and cognitive positivity). Total score is calculated from summating all items. Behavioral score is the sum or items 1-5, whereas the cognitive domain is the sum of items 6-14.

OTHER OUTCOMES:
Weight change | Baseline (week 0), immediately after the intervention (week 6)
  Weight will be measured at each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Following our extended analysis period, de-identified data will be made available, as well as the variable key, to the scientific community. Before this time, a request for data sharing will be assessed by study personnel (PI and Co-Is) as needed. These requests will be evaluated based on scientific merit and overlap with the aims of the current study.
Supporting Information: Study Protocol, SAP
Time Frame: For 5 years following final data analysis
Access Criteria: De-identified data can be made available on encrypted servers for researchers whose research plans do not overlap with the aims of the current project. Requests will be assessed by the PI and Co-Is as needed.